CLINICAL TRIAL: NCT06189131
Title: The Use of Ventriject to Assess V02Max in Patients Admitted to Hospital in the Emergency Surgery Setting
Acronym: LESS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: More funding required
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GS23/155862
Record Dates: First submitted 2023-09-26; First posted 2024-01-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Emergencies; Surgery
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups and allocation to the relevant group is based on whether the patient has required a surgical intervention during the study period. This determines which outcomes are relevant and reflects two important groups of patients admitted to emergency general surgery. The allocation to each group is finalised following completion of the data collection as the decision for operative management or conservative manage of certain pathologies can change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Acutely admitted surgical patients with no planned surgery (Experimental): This cohort of individuals will be those admitted to the EGS department with a surgical pathology but who have not undergone surgery during the admission and by the end of data collection (7 days) (e.g. pancreatitis, conservative management intra-abdominal pathology). The rationale behind recruiting this cohort of patients is to assess the admission V02Max and how unwell patients are during their admission by correlating this result to their NEWS score, blood results and any evidence of clinical deterioration. This cohort of patients will help us understand whether V02Max correlates with patient's clinical conditions and outcomes.
  Interventions: Device: Ventriject
- Group 2: Acutely admitted surgical patients who have undergone an emergency procedure (Experimental): Pre and post-operative Ventriject V02Max values will be taken in this group of patients to assess whether pre-operative V02Max correlates with pre-operative PPOSSUM, NELA scores and post-operative outcomes. This group of participants will answer whether acute V02Max is reflective of operative outcomes and whether it correlates with current methods of risk stratification (PPOSSUM, NELA, ASA) and post-operative outcome scores (Clavien-Dindo classification). This group is important as it will help establish whether V02Max measurements in the acute setting for operative risk stratification is feasible.
  Interventions: Device: Ventriject

INTERVENTIONS:
Device: Ventriject — Ventriject is a non-exercise method for estimating V02Max

SUMMARY:
The aim of this study is to assess whether Ventriject V02Max can provide values in a clinical setting and whether this value correlates with clinical outcome in patients admitted to the emergency general surgery department in a single centre. We will also be assessing the acceptability of the device to patients and clinicians.

DETAILED DESCRIPTION:
Pre-operative risk stratification is an important aspect of clinical decision-making in patients undergoing surgery. Thorough pre-operative assessment aids in the evaluation of mortality and morbidity on an individual basis and enhances the process of shared decision-making. This is particularly important in emergency surgery, which is associated with higher morbidity and mortality than elective surgery. Emergency general surgery accounts for approximately 11% of surgical cases but represents 47% of all surgical related deaths and 28% of complications. Colorectal cancer surgery has demonstrated a 90-day mortality rate of 3.2% (NBOCA 2017) and is associated with complication rates of up to 30% (Luca et al 2014). In the emergency setting, the 90-day mortality after bowel cancer surgery rises to 8.7% (NBOCA 2021).

Cardiorespiratory fitness (CRF) is an independent risk factor for mortality and morbidity for individuals undergoing surgery (Older et al, Wilson et al). Cardiorespiratory complications are the leading cause of death in non-cardiac surgery (Devereaux et al 2015, Gupta et al 2011). The insult of surgery can cause a 40% reduction in CRF for individuals with a hospital stay of up to 9 days and only half of patients regain their CRF after 6 months (Jensen et al 2011).

Cardiopulmonary exercise testing (CPET) is an exercise stress test used before planned surgery to aid risk stratification of individual patients. The CPET test involves a treadmill exercise or cycle ergometry to assess anaerobic threshold (AT) and the peak oxygen uptake (V02 peak) (Older et al 2017. CPET is a method of quantifying CRF. CPET testing is limited in certain patient populations, such as those with a physical disability or arthritis. It is time-consuming, taking approximately 40-60 minutes per assessment. A survey of patients' experiences of CPET testing was conducted by Boyd in 2016. Several aspects of CPET were described as a "serious problem" and these included dryness in mouth (11%), muscle soreness (10%), being uncomfortable (8-9%) and coughing (9%). Generally, patients requiring emergency surgery will be too unwell to preform CPET testing, but also the combination of access to facilities and the time constraints of emergency surgery make CPET testing in an emergency scenario inappropriate.

Currently there are several scoring tools used to assess a patient's risk of surgery in the emergency setting, which include PPOSSUM and NELA. These scoring tools aid in the risk stratification of mortality and morbidity to aid in the decision making for clinicians and patients. Patient characteristics integrated in these scoring tools include evidence of cardiorespiratory dysfunction assessed on ECG and clinical evidence, blood pressure, heart rate and blood test results. However, there currently is no established method of measuring CRF in the emergency setting.

Ventriject is a non-exercise method for estimating V02Max. V02Max is defined as the metabolic rate at which oxygen uptake plateaus despite further increases in work rate and this maximum end point is rarely reached during CPET examinations. V02Max has been shown to relate to post operative outcomes (Scholes et al 2009).

Ventriject uses seismocardiography (SCG) signals generated by the vibrations from a beating heart, picked up by a small accelerometer placed on the chest. SCG is an alternative method of assessing cardiac function (Sorensen et al). V02Max is estimated from the SCG signal and patient demographics including gender, age, height and weight, using machine learning. Ventriject has been tested against CEPT in over 400 healthy subjects and has been found to closely correlate with V02Max measurements (0.80, p<0.001). This is the closest correlation to ergometer testing when compared to alternative methods.

It is estimated that each Ventriject assessment costs approximately £15 and takes a total of 120 seconds to complete. It requires no physical exercise and may be more acceptable in certain clinical situations and patient groups. Currently, Ventriject has been used in non-clinical settings and lacks evidence as to its usability in the clinical environment. Given the advantages of a cheap, rapid, and accessible method of measuring V02Max, Ventriject would be an appropriate method for measuring CRF in the emergency setting and may compliment the current risk stratification tools to aid in the clinical decision making around emergency surgery.

The aim of this study is to assess whether Ventriject V02Max can provide values in a clinical setting and whether this value correlates with clinical outcome in patients admitted to the emergency general surgery department in a single centre. We will also be assessing the acceptability of the device to patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* Admitted under the General Surgery team within the last 24- 48 hours
* Anticipated hospital stay of a minimum of 48 hours

Exclusion Criteria:

Patients who are unable to consent for participation in the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-11-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
The ability for Ventriject to detect a V02Max value in individual patients | 7 days
  VO2 Max

SECONDARY OUTCOMES:
The acceptability of the device to patients | 7 days
  The acceptability of the device to patients
The correlation between V02Max with the patients NEWS score, blood results, clinical deterioration & ASA grade. Group 2: The above in addition, PPOSSUM score, NELA score, Clavien Dindo Classification | 7 days
  The correlation between V02Max with the patient clinical conditions and outcomes
The correlation between V02Max with the patients NEWS score, blood results, clinical deterioration, ASA grade, PPOSSUM score, NELA score & Clavien Dindo Classification | 7 days
  The correlation between V02Max with the patient clinical conditions and outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bautista, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lucas DJ, Pawlik TM. Quality improvement in gastrointestinal surgical oncology with American College of Surgeons National Surgical Quality Improvement Program. Surgery. 2014 Apr;155(4):593-601. doi: 10.1016/j.surg.2013.12.001. Epub 2013 Dec 14. PMID 24508118
- [Background] Jensen MB, Houborg KB, Norager CB, Henriksen MG, Laurberg S. Postoperative changes in fatigue, physical function and body composition: an analysis of the amalgamated data from five randomized trials on patients undergoing colorectal surgery. Colorectal Dis. 2011 May;13(5):588-93. doi: 10.1111/j.1463-1318.2010.02232.x. PMID 20148922
- [Background] Steffens D, Ismail H, Denehy L, Beckenkamp PR, Solomon M, Koh C, Bartyn J, Pillinger N. Preoperative Cardiopulmonary Exercise Test Associated with Postoperative Outcomes in Patients Undergoing Cancer Surgery: A Systematic Review and Meta-Analyses. Ann Surg Oncol. 2021 Nov;28(12):7120-7146. doi: 10.1245/s10434-021-10251-3. Epub 2021 Jun 8. PMID 34101066
- [Background] Scholes RL, Browning L, Sztendur EM, Denehy L. Duration of anaesthesia, type of surgery, respiratory co-morbidity, predicted VO2max and smoking predict postoperative pulmonary complications after upper abdominal surgery: an observational study. Aust J Physiother. 2009;55(3):191-8. doi: 10.1016/s0004-9514(09)70081-9. PMID 19681741
- [Background] Wilson RJ, Davies S, Yates D, Redman J, Stone M. Impaired functional capacity is associated with all-cause mortality after major elective intra-abdominal surgery. Br J Anaesth. 2010 Sep;105(3):297-303. doi: 10.1093/bja/aeq128. Epub 2010 Jun 23. PMID 20573634
- [Background] Older P, Smith R, Courtney P, Hone R. Preoperative evaluation of cardiac failure and ischemia in elderly patients by cardiopulmonary exercise testing. Chest. 1993 Sep;104(3):701-4. doi: 10.1378/chest.104.3.701. PMID 8365279
- [Background] Sorensen K, Schmidt SE, Jensen AS, Sogaard P, Struijk JJ. Definition of Fiducial Points in the Normal Seismocardiogram. Sci Rep. 2018 Oct 18;8(1):15455. doi: 10.1038/s41598-018-33675-6. PMID 30337579
- [Background] Devereaux PJ, Sessler DI. Cardiac Complications in Patients Undergoing Major Noncardiac Surgery. N Engl J Med. 2015 Dec 3;373(23):2258-69. doi: 10.1056/NEJMra1502824. No abstract available. PMID 26630144
- [Background] Gupta H, Gupta PK, Fang X, Miller WJ, Cemaj S, Forse RA, Morrow LE. Development and validation of a risk calculator predicting postoperative respiratory failure. Chest. 2011 Nov;140(5):1207-1215. doi: 10.1378/chest.11-0466. Epub 2011 Jul 14. PMID 21757571
- See also: national-bowel-cancer-audit-annual-report-2017 — http://www.hqip.org.uk/resource/national-bowel-cancer-audit-annual-report-2017